CLINICAL TRIAL: NCT06147492
Title: Urinary Retention Following Transanal Versus Laparoscopic Total Mesorectal Excision for Rectal Cancer
Brief Title: Urinary Retention Following taTME VS laTME Total Mesorectal Excision for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Director, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIH-SYip66
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: urinary retention
MeSH Terms: conditions — Rectal Neoplasms; Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laTME (Other): Laparoscopic Total Mesorectal Excision
  Interventions: Procedure: Laparoscopic Total Mesorectal Excision
- taTME (Other): a transanal bottom-up approach was employed for the Total Mesorectal Excision procedure
  Interventions: Procedure: transanal total mesorectal excision; Procedure: Laparoscopic Total Mesorectal Excision

INTERVENTIONS:
Procedure: transanal total mesorectal excision — a transanal bottom-up approach was employed for the TME procedure
  Arms: taTME
Procedure: Laparoscopic Total Mesorectal Excision — Laparoscopic Total Mesorectal Excision

SUMMARY:
A comprehensive study with prospectively collected data. These patients were assigned to either the taTME group or the laTME group according to the surgery procedure received

DETAILED DESCRIPTION:
Transanal total mesorectal excision has emerged as a potential solution to certain limitations associated with laparoscopic total mesorectal excision in rectal cancer patients. Differences in surgical approaches have raised questions regarding their impact on the risk of postoperative urinary retention, with limited data available from large scale study.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 65 years,
* Diagnosed with rectal cancer at clinical tumor node metastasis stages II or III.
* Palpable tumor determined by digital rectal examination or proctoscopy
* The distal border of the tumor located within 12 cm from the anal verge

Exclusion Criteria:

* Patients presenting clear indications of pelvic side wall involvement or distant metastasis
* Uncontrolled hypertension or cardiovascular disease
* Patients with synchronous colon cancer
* History of other malignancies within the past 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
urinary retention | 30 days
  urinary retention rate

IPD SHARING:
Plan to Share IPD: No
upon reasonable request